CLINICAL TRIAL: NCT07333703
Title: MRI-Based Estimation of Lumbar CSF Volume and Its Clinical Impact on Spinal Anaesthesia
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: SUKAEK-2022/1/14
Record Dates: First submitted 2025-11-21; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Spinal Anaesthesia; Magnetic Resonance Imaging (MRI); Lumbosacral Spinal Stenosis; Anaesthesia
Keywords: Spinal Anaesthesia; Peak sensory block level; Lumbosacral volume; MRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Distribution of spinal anesthetic agent — Under aseptic conditions and in a sitting position, a 25G spinal needle was inserted through the midline at the L₃-L₄ intervertebral space, advancing parallel to the dura fibers. Upon clear cerebrospinal fluid (CSF) flow, the needle bevel was oriented cephalad and 20 mg of 0.5% hyperbaric bupivacaine was injected into the intrathecal space. Patients were kept supine for 5 minutes before sensory block was assessed by pinprick test from the midclavicular line. All spinal anesthesia procedures were performed by the same experienced anesthesiologist.

SUMMARY:
This prospective observational study aims to investigate the clinical impact of lumbar cerebrospinal fluid (CSF) volume on spinal anesthesia characteristics. A total of 40 adult patients, aged 18 to 75 years and classified as ASA physical status I-III, who had undergone 3D T2-weighted lumbosacral MRI within the past six months, were enrolled. Intrathecal anesthesia was administered with 4 mL (20 mg) of 0.5% hyperbaric bupivacaine via the L3-L4 interspace in a sitting position.

CSF volume was measured from the lower half of the L1 vertebral body to the sacral end using the volume of interest (VOI) method on sagittal 3D T2-weighted MR images, processed with the ITK-SNAP software. Primary outcome was the correlation between lumbosacral CSF volume and peak sensory block level. Secondary outcomes included correlations with the onset time and duration of sensory and motor block, two-segment regression time, and patient characteristics such as height, weight, BMI, and age.

DETAILED DESCRIPTION:
Spinal anesthesia is a widely used and effective alternative to general anesthesia for surgeries performed below the L₁-L₂ level, where the spinal cord ends. However, the distribution and duration of local anesthetics in spinal anesthesia are often unpredictable due to factors such as anesthetic dose, injection speed and location, patient position, age, and body habitus. One important yet less predictable factor is the individual variability in cerebrospinal fluid (CSF) volume, especially in the lumbosacral region. Since CSF dilutes the intrathecally administered anesthetic, differences in CSF volume can significantly impact drug concentration and, consequently, block level and duration.

Advancements in imaging techniques such as ultrasound and MRI have contributed to more accurate estimations of CSF volume. While most studies have used ultrasound-based estimations, MRI-based evaluations remain limited. In this study, we aimed to investigate the effect of lumbosacral CSF volume, measured via 3D T₂-weighted MRI, on the duration and extent of spinal anesthesia. Understanding this relationship could improve predictability in spinal anesthesia and enhance personalized anesthetic planning.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years
* ASA physical status I-III
* Who had undergone 1.5 Tesla lumbosacral MRI within the last six months

Exclusion Criteria:

* The presence of neurological diseases and allergy to local anesthetics
* Refusal to undergo spinal anesthesia
* Contraindications for spinal anesthesia
* Local infection at the lumbar site

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged between 18 and 75 years, classified as ASA physical status I-III, who had undergone 1.5 Tesla lumbosacral MRI within the last six months.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
The primary outcome was to assess the correlation between lumbosacral CSF volume and peak sensory block level. | From enrollment to the end of study 33 months

CONTACTS AND LOCATIONS:
Locations (1):
- Samsun University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stienstra R, Greene NM. Factors affecting the subarachnoid spread of local anesthetic solutions. Reg Anesth. 1991 Jan-Feb;16(1):1-6. No abstract available. PMID 2007097